CLINICAL TRIAL: NCT02912000
Title: TEACH: Technology Evaluation to Address Child Health
Acronym: TEACH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Academic Pediatric Association (Industry); Fonds de la Recherche en Santé du Québec (Other Government)
Responsible Party: Principal Investigator, Jonathan P. Winickoff, MD, MPH, MD, Massachusetts General Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2016P000711/MGH
Record Dates: First submitted 2016-09-21; First posted 2016-09-23 (Estimated); Last update posted 2018-03-22 (Actual); Status verified 2018-03

CONDITIONS: Smoking; Obesity; Dental Caries
Keywords: Dental Health Services; Sugar-Sweetened Beverages; Tobacco control; Pediatrics; Parents
MeSH Terms: conditions — Smoking; Obesity; Dental Caries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Experimental): The intervention group will receive the TEACH intervention - an electronic tablet screening in waiting room for the modifiable risk factors
  Interventions: Behavioral: TEACH intervention
- Control (No Intervention): Care as usual: No electronic tablet in waiting room

INTERVENTIONS:
Behavioral: TEACH intervention — The TEACH intervention screens family for three modifiable behaviors ahead of the clinical encounter: parental tobacco use, children consumption of sugar-sweetened beverages and child dental health. The information from the screening is then shared with clinicians.
  Arms: Intervention

SUMMARY:
The proposed study is a pre- /post-implementation study in a pediatric practice with a control practice designed to test the feasibility and effectiveness of an electronic screening and service delivery tool for three modifiable health risk factors in pediatrics: parental tobacco use, sugar-sweetened beverages consumption, and poor dental care

DETAILED DESCRIPTION:
Key procedures of the study include:

1. Practices will be contacted via letters, emails and in-person discussion with practice leaders.
2. Among practices that say yes to recruitment, a total of 2 practices will be randomly assigned to one of two groups: 1) Implementation of the electronic screening tool 2) care as usual
3. Control and intervention practices will be trained in integrating a Research Assistant (RA) who will be hired, trained, and paid by the research study. RAs will be through networking, temporary officeservice contractors, and other local resources.
4. A notice to parents and teenagers will be posted where all can see it when registering for their pediatric visit. The notice will announce that the practice is participating in a research study and that parents/guardians and teenagers may be approached by a study RA. Practice staff will refer parents to the RA for the Eligibility Screener.
5. In the control practice and in the pre-implementation phase of the intervention practice, after being seen by the pediatric clinician, the parent will be approached by the RA stationed near the exit of the clinic for an exit interview consisting of the Exit Survey. Alternatively, it the practice prefers to not have RAs directly approaching patients, practice staff will refer the potential participants to the RA after checkout. Parents who agree to study participation will learn about the study, sign the consent, and complete the Exit Survey for enrolled parents/guardians. Teenagers will not be invited or involved in this part of the study.
6. In the post-implementation phase of the intervention practice, practice staff will follow a script at the check-in desk to refer parents to the RA. Parents will be approached by the RA after checking in for their appointment. Parents who agree to study participation will complete the Intake Survey. If they are accompanied by a teenager (aged 13-18 years old, the teenager will also be presented the study. Parents will be invited to consent to their child participate in the study. If the child is 13 years old, we will seek assent from the child to answer a portion of the intake survey. If he/she is 14 years or older, consent will be sought, and if obtained, the teenager will be asked to complete a section of the survey, on the same risk factors. We are asking that written documentation of these being waived and that consent/assent be inferred from survey participation, which will be documented in the research record. Teenagers will not be compensated for this section of the study that should take less than 5 minutes to complete. After completion of the survey, the adult participants will receive, if they desire, an information sheet on the risk factors identified, as well as a summary of the screening questionnaire, to be handed to the clinician they are coming to see that day. If no risk factor is identified, no clinician handout will be given. Teenagers' response to the survey will not be shared with parents and will only be available to the principal investigator and co-investigator. Adult participants will also be asked to reach out to the RA after their appointment to complete the Exit Survey, following the procedure mentioned above.
7. One month after the recruitment and completion of the Exit Survey, adult participants will be contacted by phone by the RA or the Principal Investigator (PI) to complete the Follow-up survey. Consent for this survey will be obtain as part of the study initial consent and preferred phone numbers will be obtained directly from the participants. After completion of the Follow-up Survey, participation in the survey will be complete.

ELIGIBILITY:
Inclusion Criteria:

* Parent of a child aged 0-18 years

Exclusion Criteria:

* Parents under age 18
* Parents who have a child with a medical emergency (any condition requiring transfer for immediate medical intervention)
* Non-consenting individuals
* Non-English speakers

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 650 (Actual)
Dates: Start 2016-09; Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Reported screening and counseling by physicians about parental smoking, child dentist appointment, and sugar-sweetened beverages | Pre-implementation (baseline) and Post-implementation
  Higher rates of screening, counseling, and service delivery by clinicians in the period after implementation than at baseline (pre-implementation).

SECONDARY OUTCOMES:
Parent report of behavior change intention related to parental smoking, child sugar sweetened beverage consumption and child's dental appointment | At baseline and one month follow-up
  Compared to the pre-implementation period, parents in the post-implementation period will have greater behavior change intention for each modifiable risk factor. This difference will be greater in the intervention practice than in the control practice.
Reported behavior change related to parental smoking, child sugar sweetened beverage consumption and child's dental appointment | one month follow-up
  At one month follow-up, the intervention group will have a greater increase in reported healthy behavior than the control group.

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan P Winickoff, MD MPH, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided